CLINICAL TRIAL: NCT05116553
Title: Motivational Evaluation and Intervention With Co-Adapt Application for Healthy Ageing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Idego srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COADAPT 2021 T-6.4
Record Dates: First submitted 2021-10-26; First posted 2021-11-11 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Motivation; Self Efficacy
Keywords: Motivation; Self efficacy

STUDY DESIGN:
Intervention Model Description: Pre-intervention test will be administered to the participants (T1) to assess their psychological well-being, motivation, awareness of change, self-confidence and self-efficacy.
  Participants will be randomly divided into two group: the experimental group will receive the standard 2 Self Determination Theory (SDT) psychological interviews with the support of the APP with the Conversational Agent (CA), while the control group will receive the 2 SDT (Self Determination Theory) psychological interviews.
  At the end of the pathway post-intervention test (T2) will be administered to the participants with the same questionnaire of the beginning.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDT (MI) (Active Comparator): This group will receive standard 2 SDT (Self Determination Theory) psychological interviews.
  Interventions: Behavioral: SDT
- SDT (MI) + CA (Experimental): This group will receive standard 2 SDT (Self Determination Theory) psychological interviews; moreover they will use an APP with a CA (Conversational Agent), an Artificial Intelligence.
  Interventions: Behavioral: SDT; Device: APP + CA

INTERVENTIONS:
Behavioral: SDT — Standard 2 SDT (Self Determination Theory) psychological interviews.
Device: APP + CA — An APP with a CA (Conversational Agent).
  Arms: SDT (MI) + CA

SUMMARY:
The aim of this study is to identify effective methodologies to help people to improve their awareness of change, motivation, self-confidence and self-efficacy, compliance in behavioral change and psychological well-being.

DETAILED DESCRIPTION:
Subjects involved will have the opportunity to partecipate in a two-weeks course: two SDT (Self Determination Theory) psychological interviews are scheduled (1 per week) to help the participant increase his motivation and awareness about the problem reported during the counseling session.

For this purpose, the use of an APP with a CA (Conversational Agent) will be implemented as a support to help people to identify one's thoughts and emotional states as well as increase their awareness about themselves.

Test will be administered at the beginning (T1) and at the end of the meetings (T2).

Participants will be randomly divided into one of two groups to understand whether APP and CA has a significant impact in increasing motivation and awareness of the need for a pathway with a professional.

ELIGIBILITY:
Inclusion Criteria:

* whitecollar
* a sufficient level of education to understand study procedures and be able to communicate with site personnel
* 50 to 70 years old

Exclusion Criteria:

- current use of narcotics or other substances

Ages: 50 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Change in levels of General Self-Efficacy Scale-10 (GSE-10) | Up to day 14
  GSE-10 test is a validated test for the detection of general self efficacy. The total score ranges from 10 to 40. Higher scores mean better outcomes.
Change in levels of Basic Psychological Need Satisfaction and Frustration Scale (BPNSFS) | Up to day 14
  The BPNSFP-24 test is a validated test for the detection of the satisfaction and frustration of the primary needs: autonomy, relatedness and competence (according to SDT Theory). The total score ranges from 24 to 120. Higher scores mean better outcomes.

SECONDARY OUTCOMES:
Change of the scales contained in the Depression Anxiety Stress Scales-21 (DASS-21) | Up to day 14
  The DASS-21 test is a validated test for the detection of depression, anxiety and stress. The total score of each subscale ranges from 0 to 42. Higher scores mean worse outcomes.
Change in World Health Organisation-Five Well-Being Index (WHO-5) | Up to day 14
  The WHO-5 test is a validated test for the detection of psychological wellbeing. The total score ranges from 0 to 100. Higher scores mean better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Ciulli, Principal Investigator — Idego srl
Locations (1):
- Idego srl, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Clinical data obtained from psychological testing and socio-demographic data and any feedback collected during the trial will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available starting in February 2022
Access Criteria: The data available on the research website (www.co-adapt.it). A special page will be created where researchers can download the raw data to perform any analysis.